CLINICAL TRIAL: NCT00422994
Title: An Open-Label, Parallel-Group, Repeat-Dose Study to Investigate the Effects of End Stage Renal Disease and Haemodialysis on the Pharmacokinetics of Ropinirole (Study RRL103628)
Brief Title: A Study To Investigate The Effects Of End Stage Renal Disease And Hemodialysis On The Pharmacokinetics Of Ropinirole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RRL103628
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome
Keywords: end stage renal impairment; tolerability; ropinirole; pharmacokinetics; hemodialysis
MeSH Terms: conditions — Restless Legs Syndrome

INTERVENTIONS:
Drug: ropinirole dosing for up to 28 days

SUMMARY:
This study will investigate the effects of severe renal impairment and hemodialysis on the characteristics of the drug, ropinirole.

ELIGIBILITY:
Inclusion:

* Patients and subjects between 18-79 years old.
* End stage renal patients who are consistently receiving dialysis for a minimum of 3.5 hours, three times per week, with hemodialysis blood flow rates of >200mL/min may be eligible to enter the study.
* Patients must also have systolic blood pressure 100-190mmHg and diastolic blood pressure <120mmHg.
* Healthy subjects must have systolic blood pressure 100-150mmHg.

Exclusion:

* Female subjects who are pregnant and/or breast-feeding must not participate in this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
SK&F-104557 and SK&F-89124 blood levels over 24 hours at Weeks 1 & 3 for all subjects.
SK&F-104557 and SK&F-89124 blood levels at beginning, middle, & end of hemodialysis period when "on dialysis" & "off dialysis" in patients.

SECONDARY OUTCOMES:
ECG: every other visit
Vital Signs: Each visit
Adverse Events: each visit
Clinical laboratory: every other visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Minneapolis, Minnesota, United States
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: RRL103628 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register